CLINICAL TRIAL: NCT06289400
Title: Investigating the Effect of Magnetic Field Application Used in Patellofemoral Pain Syndrome
Brief Title: Magnetic Field Application in Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUOAS
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-02

CONDITIONS: Pain, Knee
Keywords: Pain, Knee, Magnetic field, Physiotherapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Conventional treatment+ Magnetic field application
  Interventions: Device: Magnetic field application; Other: Conventional treatment
- Control Group (Active Comparator): Conventional treatment
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: Magnetic field application — The applicator (Size: 15x15 cm) has placed 1-3 cm above the skin surface at the painful area. During the treatment, treatment has applied with ready-made protocols included in the device.
  Arms: Study Group
Other: Conventional treatment — Within the scope of conventional treatment, hotpack application, transcutaneous electrical stimulation (TENS), interferential current and ultrasound treatment modalities will be applied. In addition, strengthening exercises will be applied to the muscles around the hip and knee and stretching exercises will be applied to the short muscle groups.

SUMMARY:
The purpose of this study is to examine the effect of magnetic field application used in the treatment of patellofemoral pain.

DETAILED DESCRIPTION:
The aim of this randomized controlled study is to examine the effect of magnetic field application used in the treatment of patellofemoral pain.

The main question it aims to answer is;

Is magnetic field therapy applied in addition to conventional treatment effective in reducing pain in individuals with Patellofemoral pain syndrome?

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with patellofemoral pain syndrome by an orthopedic physician
* Volunteering to participate in the study
* Having pain for more than eight weeks
* Patients who did not undergo surgery

Exclusion Criteria:

* Patients diagnosed with rheumatological disease
* Patients who have previously had steroid injections in the knee area
* Patients with entrapment neuropathy and deformity in the lower extremity
* Patients who are pregnant
* Patients suffering from scoliosis,
* Patients who use non-steroidal anti-inflammatory and antidepressant regularly for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | The evaluation will be applied at the beginning of the treatment program.
  A Visual Analogue Scale (VAS) is one of the pain rating scales.Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.
36-Item Short Form Survey (SF-36) | The evaluation will be applied at the beginning of the treatment program.
  The SF-36 is a 36-item self-report measure of health-related quality of life. It has eight subscales measuring different domains of health-related quality of life: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH).
Manual Muscle Test | The evaluation will be applied at the beginning of the treatment program.
  Manual muscle testing is based on the physiotherapist manually applying resistance to the muscle or muscle group to be evaluated.
The Lower Extremity Functional Scale (LEFS) | The evaluation will be applied at the beginning of the treatment program.
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Karaca, PhD, Study Chair — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)